CLINICAL TRIAL: NCT04540003
Title: School Based Health Care: A Model for Improving Educational Achievement for Children in Inner City Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Toronto District School Board (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-341
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Educational Achievement
Keywords: school-based health centre; SBHC; School Support Team; SST; academic; inner city schools; standardized test scores; developmental pediatrics; education; achievement

STUDY DESIGN:
Intervention Model Description: This project will be a prospective cohort quasi-experimental study design to compare the benefits of using SBHCs as opposed to the traditional health care by evaluating educational achievements. The study period includes September 2017-June 2018 and September 2018-June 2019. Of 16 inner city schools not previously exposed to the SBHC in the TDSB, some schools (n=8) will be in the control arm following the standard of care while others (n=8) will have access to SBHC. Students presented to SST meetings whose outcomes include the need for a developmental/pediatric assessment at the 16 schools will be identified by TDSB internal research staff. To conduct our primary analysis, standardized test scores and numeric data from report cards will be analyzed using a linear mixed effect model where the schools are the random effects and the baseline test scores and report cards are adjusted for by including it as a covariate.
Masking Description: It is not feasible to blind students or their families or SST members as there are obvious differences in care procedures between the two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to School Based Health Centre (Experimental): Of the eight school in the intervention arm, four schools will be linked to a school based health center (SBHC) at Sprucecourt or Nelson Mandela Park Public Schools (established in partnership with the department of Pediatrics at St. Michael's hospital) and four schools will be linked to a SBHC at Parkdale Public School (established in partnership with St. Joseph's Health Centre). SBHC pediatricians will attend School Support Team (SST) meetings at all intervention schools and students with developmental concerns identified at the SST meetings will be referred to the SBHC.
  Interventions: Other: Access to School Based Health Centre
- Control Arm: Standard of care (No Intervention): Of the eight schools assigned to the control condition, four will be in the South East area of the city closer to Nelson Mandela Park PS and four will be in the South West area of the city closer to St. Josephs Health Center. The eight schools will be subject to standard of care which is: when a child is identified by the SST (no pediatrician present), students identified with developmental concerns are advised to access a pediatric/developmental assessment in the community.

INTERVENTIONS:
Other: Access to School Based Health Centre — The SBHC will be staffed by a family physician, two pediatricians and a developmental pediatrician, each with at least one half-day of clinic time per week from September through June. The SBHC is also staffed by a clinic coordinator who is responsible for booking appointments on a first-referral, first-serve basis.
  Arms: Access to School Based Health Centre

SUMMARY:
Developmental problems have tremendous impact on children, affecting academic achievement and mental health later in life.The process of receiving a developmental assessment is long and arduous, and may require multiple physician visits taking over one year. Although a relatively new concept in Canada, School-Based Health Centres (SBHCs) have been successfully implemented in over 1900 schools in the United States.The first SBHC in Ontario, and Canada as a whole, was established through the Model Schools Pediatric Health Initiative (MSPHI) and is dedicated to reducing health inequities for inner city children by reducing barriers and providing accessible clinical care. To provide more conclusive evidence on the relative benefits of SBHCs as compared to traditional health care access, this study will use a prospective cohort quasi-experimental study design to compare differences in educational achievement for developmental assessments in the SBHC model relative to standard care. As per standard of care, students having difficulty in school are identified by the Toronto District School Board (TDSB) internal research staff and are presented to the monthly School Support team (SST) meetings. Historically physicians do not attend SST meetings, however, as a part of the SBHC program, pediatricians will participate in monthly SST meetings. Schools assigned to the intervention group will have SBHC physicians attend SST meetings, while schools assigned to the control group will not.

The overall objective of this study is to examine educational achievement, as defined by standardized test scores and report cards in students who use an inner city SBHCs for developmental concerns relative to those who do not. We hypothesize students attending schools in which SST meetings have a pediatrician present, that are referred to a SBHC, will score higher and show a greater increase in standardized test scores and report cards (from baseline to follow-up) than students attending schools in which SST meetings do not have a pediatrician present and access services through traditional means in the community (standard of care).The secondary objectives are: a) to examine socio-demographic data for these students and its relationship to educational achievement and b) to determine wait times to developmental assessment for students in the intervention group who attend the SBHCs using retrospective chart review.

ELIGIBILITY:
Inclusion Criteria:

* All students identified at the SST meetings requiring a developmental assessment.

Exclusion Criteria:

* Students without a developmental concern and not identified at the SST meeting will be excluded. No other specific exclusion criteria will be applied.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Educational achievement as assessed by numeric data from report cards. | Change from baseline to 18 months after identification at SST
  For each student attending the schools enrolled in this study, the report cards have the student's grade for all the core subjects reported as a percentage (0-100%). The higher the grade the better the academic performance. There is also the class median reported as a percentage so that the student's academic performance in that particular subject can be compared to that of their class's average performance for that same subject.
  Numeric data from report cards will be analyzed using a linear mixed effect model where the schools are the random effects and the baseline report cards are adjusted for by including it as a covariate. Baseline report cards will be determined as those that have occurred most proximal to the SST date. The treatment effect will be expressed as the mean adjusted difference in standardized test scores with 95% confidence interval.
Educational achievement as assessed by Canadian Achievement Test 4 (CAT4) scores. | Change from baseline to 18 months after identification at SST
  The Canadian Achievement Test 4 (CAT4) is a standardized test administered to students in grades 1-6 across Canada to assess basic skill areas: reading, writing, and mathematics. Higher scores mean better outcome. The raw score (0-100%) on each test section is converted to a national stanine range (1-9), where scores in the range of 1-3 is considered below-average (i.e. Low (L)), scores in the range of 4-6 are considered average (i.e. Competent (C)) and scores 7-9 are considered above average (i.e. Proficient (P)) performence.
  Standardized test scores will be analyzed using a linear mixed effect model where the schools are the random effects and the baseline test scores are adjusted for by including it as a covariate. Baseline test scores will be determined as those that have occurred most proximal to the SST date.The treatment effect will be expressed as the mean adjusted difference in standardized test scores with 95% confidence interval.
Education achievement as assessed by Education Quality and Accountability Office (EQAO) scores | Change from baseline to 18 months after identification at SST
  Toronto District School Board (TDSB) Standardized tests include the Education Quality and Accountability Office (EQAO) test. The EQAO is a test that assesses literacy and math skills and is administered to students in grades 3 and 6. Based on the student's performance on the EQAO, the student's raw score is converted into a score on a scale from 200 (level 2) to 400 points (level 4). A score of 300 (level 3) (i.e. average student score) is required to be successful. A score above 300 (i.e. level 4 (400 points)) is considered above average.
  Standardized test scores will be analyzed using a linear mixed effect model where the schools are the random effects and the baseline test scores are adjusted for by including it as a covariate. Baseline test scores will be determined as those that have occurred most proximal to the SST date.The treatment effect will be expressed as the mean adjusted difference in standardized test scores with 95% confidence interval.

SECONDARY OUTCOMES:
Socio-demographic data and relationships to educational achievement | change from baseline to 18 months after identification at SST
  Children from inner city schools may face additional difficulties accessing healthcare to address developmental and mental health concerns, particularly when they come from families with socioeconomic challenges, language barriers and limited means of transportation. Data collection will entail the collection of in-depth, in-person interviews with each participant 18 months after the SST meeting in both arms. During baseline interviews, participants will be asked questions regarding their current experiences (and contexts) at the outset of the trial. At the end of the trial, participants will be asked to reflect on their experiences before the trial began, how their experiences and perspectives changed as a result of the trial, and their reflections on trial implementation. Interviews will be conducted by experienced qualitative research personnel, audio taped and transcribed verbatim.
Wait time data will be determined retrospectively from chart review for the intervention group | date of SST meeting to date of developmental assessment
  Charts of students attending the SBHC from the schools in the intervention arm will assessed for the following only: date of SST meeting, date of first visit to SBHC, date of developmental assessment. This will be used to determine the wait time. Wait times will be reported as a mean and standard deviation. Since data from the TDSB is de-identified, we will not be linking wait time data with outcomes or any other data provided by the TDSB.

CONTACTS AND LOCATIONS:
Overall Officials: Sloane Freeman, MSc,MD,FRCPC, Principal Investigator — Unity Health Toronto
Locations (1):
- Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Breslau J, Miller E, Breslau N, Bohnert K, Lucia V, Schweitzer J. The impact of early behavior disturbances on academic achievement in high school. Pediatrics. 2009 Jun;123(6):1472-6. doi: 10.1542/peds.2008-1406. PMID 19482756
- [Background] Reynolds AJ, Temple JA, Ou SR, Robertson DL, Mersky JP, Topitzes JW, Niles MD. Effects of a school-based, early childhood intervention on adult health and well-being: a 19-year follow-up of low-income families. Arch Pediatr Adolesc Med. 2007 Aug;161(8):730-9. doi: 10.1001/archpedi.161.8.730. PMID 17679653
- [Background] Shevell MI, Majnemer A, Rosenbaum P, Abrahamowicz M. Profile of referrals for early childhood developmental delay to ambulatory subspecialty clinics. J Child Neurol. 2001 Sep;16(9):645-50. doi: 10.1177/088307380101600904. PMID 11575603
- [Derived] Rasiah S, Juni P, Sgro MD, Thorpe KE, Maguire J, Freeman SJ. School-based health care: improving academic outcomes for inner-city children-a prospective cohort quasi-experimental study. Pediatr Res. 2023 Oct;94(4):1488-1495. doi: 10.1038/s41390-023-02473-w. Epub 2023 Feb 8. PMID 36755187